CLINICAL TRIAL: NCT07260695
Title: Study Evaluating Visual Outcomes in Post-Myopic LASIK Patients After Implantation of the Odyssey Intraocular Lens
Brief Title: Odyssey Evaluation in Post LASIK Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Center For Sight (Other)
Collaborators: Sengi Clinical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFS 25-001
Record Dates: First submitted 2025-08-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Odyssey IOL (Other)
  Interventions: Device: Odyssey intraocular lens

INTERVENTIONS:
Device: Odyssey intraocular lens — The Odyssey intraocular lens is intended to be implanted at the time of cataract surgery to replace the natural lens.

SUMMARY:
This prospective study evaluates the visual and refractive outcomes of the TECNIS Odyssey intraocular lens (IOL) implanted in patients with a history of myopic LASIK. Given the unique optical challenges of post-LASIK eyes, including altered corneal curvature and higher-order aberrations, the study aims to assess the IOL's performance in terms of distance, intermediate, and near vision, and patient satisfaction. Its design features may offer favorable outcomes in these patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST fulfill the following conditions to qualify for enrollment into the trial

1. Age: 50 years and older.
2. Gender: Males and Females.
3. Bilateral cataracts
4. Bilateral implantation of Odyssey IOLs (toric and non-toric)
5. Scheduled to undergo standard cataract surgery in both eyes, within 1 to 30 days between surgeries.
6. Willing and able to provide written informed consent for participation in the study.
7. Willing and able to comply with scheduled visits and study examination procedures.
8. Postoperative best corrected visual acuity of 0.2 logMAR (20/32 Snellen) or better in each eye.

Exclusion Criteria:

Subjects with ANY of the following conditions on the eligibility exam may NOT be enrolled into the trial.

1. Established ocular pathology, including: glaucoma (except glaucoma suspects), uveitis, and clinically-significant retinal pathology affecting the macula (with visual acuity worse than 20/25) and/or any other ocular findings that may, in the opinion of the investigator, affect vision.
2. Uncontrolled diabetes.
3. Use of any systemic or topical drug known to interfere with visual performance.
4. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
5. Clinically significant corneal dystrophy.
6. Contact lens use during the active treatment portion of the trial.
7. Irregular astigmatism.
8. Corneal irregularities potentially affecting visual acuity (i.e., keratoconus, corneal opacities
9. History of chronic intraocular inflammation.
10. History of retinal detachment.
11. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
12. Previous intraocular surgery.
13. Previous keratoplasty
14. Previous refractive surgery other than myopic LASIK or PRK (i.e., radial keratotomy, hyperopic LASIK, etc)
15. Severe dry eye.
16. Pupil abnormalities.
17. Subject who may reasonably be expected to require a secondary surgical intervention at any time during the study (other than YAG capsulotomy, i.e., LASIK).
18. Any clinically significant, serious, or severe medical or psychiatric condition that may interfere with the interpretation of study results.
19. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.
20. Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
21. Abnormal iris

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates the patient is unsuitable for the trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Binocular defocus curve | 3 months postoperatively
  The defocus curve assesses a patient's visual performance at various distances by introducing different levels of lens defocus (measured in diopters) and recording the corresponding visual acuity. It provides a comprehensive evaluation of the range of clear vision (distance, intermediate, and near) offered by an intraocular lens.

SECONDARY OUTCOMES:
Patient satisfaction | 3 months postoperatively
  Percentage of patients who reported being completely, mostly, moderately, a little or not at all satisfied with overall vision
Spectacle independence at near. | 3 months postoperatively
  Percentage of patients who reported wearing glasses none of the time or a little of the time for near activities (16 inches/40 cm).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin K De Rojas, MD, Principal Investigator — Center For Sight
Locations (1):
- Center For Sight, Venice, Florida, United States

IPD SHARING:
Plan to Share IPD: No